CLINICAL TRIAL: NCT00106418
Title: An Exploratory Phase II, Multicenter, Open-label Trial Evaluating the Activity and Tolerability of FK228 in Androgen Independent Metastatic Prostate Cancer Patients With Rising PSA
Brief Title: A Research Study for Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ-228-0002; NCT00058643 (obsolete NCT alias)
Record Dates: First submitted 2005-03-24; First posted 2005-03-25 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer; Metastases
Keywords: Prostate Cancer; Androgen independent metastatic prostate cancer patients with rising PSA; romidepsin
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — romidepsin; Depsipeptides

ARMS (1):
- Romidepsin (Experimental): 13 mg/m^2 of romidepsin intravenously over 4 hours on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: Romidepsin

INTERVENTIONS:
Drug: Romidepsin — 13 mg/m2 of romidepsin intravenously over 4 hours on Days 1, 8, and 15 of each 28-day cycle.
  Other Names: Istodax; depsipeptide; FK 228

SUMMARY:
The purpose of this study is to evaluate the activity of romidepsin (depsipeptide,FK228) in patients with metastatic prostate cancer who have developed a rising prostate specific antigen (PSA) while undergoing hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥18 years;
* Written informed consent/authorization;
* Histological or cytological confirmation of metastatic prostate cancer with documented progression on hormonal therapy (objective progressive disease [PD], new bone lesions, or stable soft tissue or bone lesions with PSA increase);
* Patients must have either measurable disease or bone metastasis. Patients with measurable disease are preferred;
* Rising PSA, with a minimum study entry PSA of ≥5 ng/mL;
* Karnofsky performance status of ≥80%;
* Life expectancy of >12 weeks;
* For patients treated with anti-androgens, elevation of PSA must be demonstrated after cessation of anti-androgen treatment;
* Three lines of hormonal therapy are permitted prior to study entry (anti-androgen withdrawal is not considered as a second hormonal treatment);
* Serum testosterone level of <50 ng/mL in patients without surgical castration;
* Patients must have serum potassium levels >4.0 mEq/L and serum magnesium levels >2.0 mg/dL.

Exclusion Criteria:

* Concomitant use of any anti-cancer therapy, except for continued use of luteinizing hormone-releasing hormone (LHRH) agonists or antiandrogens, or bisphosphonates or steroids initiated at least 4 weeks prior to study entry;
* Concomitant use of any investigational agent, including PC-SPES;
* Use of any investigational agent within 4 weeks of study entry;
* Concomitant use of warfarin (due to a potential drug-to-drug interaction with depsipeptide);
* Major surgery within 2 weeks of study entry;
* Prior treatment with chemotherapy;
* Patients with known cardiac abnormalities such as:
* Congenital long QT syndrome;
* QTc interval > 480 milliseconds;
* Patients who have had a myocardial infarction within 12 months of study entry;
* Patients who have a history of coronary artery disease (CAD) e.g., angina Canadian Class II IV (see Appendix K). In any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
* Patients with an ECG recorded at screening showing evidence of cardiac ischemia (ST depression of ≥2 mm). If in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
* Patients with congestive heart failure that meets NYHA Class II to IV (see Appendix J) definitions and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or magnetic resonance imaging (MRI);
* Patients with a history of sustained VT, VF, Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
* Patients with hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other causes (in doubt, see ejection fraction criteria above);
* Patients with uncontrolled hypertension i.e., ≥160/95;
* Patients with any cardiac arrhythmia requiring anti-arrhythmic medication;
* Concomitant use of medications which may cause a prolongation of QT/QTc (see Appendix D) interval;
* Concomitant use of medications that are inhibitors of the cytochrome P-450 isoenzyme CYP 3A4 (see Appendix E);
* Clinically significant active infection;
* Known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C;
* Previous extensive radiotherapy involving 30% of bone marrow (e.g., whole of pelvis, half of spine);
* Clinical or radiological imaging evidence of brain metastasis (computed tomography [CT] or MRI scans are required only if brain metastasis is suspected clinically);
* Inadequate bone marrow or other organ function, as evidenced by:

  * hemoglobin <9.0 g/dL (transfusions and/or erythropoietin are permitted);
  * absolute neutrophil count (ANC) ≤1.5 x 109 cells/L;
  * platelet count <100 x 109 cells/L;
  * total bilirubin >1.25 x upper limit of normal (ULN) for institution or >2.0 x ULN in the presence of demonstrable liver metastases;
  * aspartate transaminase/serum glutamic oxaloacetic transaminase (AST/SGOT) and alanine transaminase/serum glutamic pyruvic transaminase (ALT/SGPT) >2.0 x ULN or >5.0 x ULN in the presence of demonstrable liver metastases;
  * serum creatinine >2 mg/dL;
* Serum potassium levels < 4.0 mEq/L and serum magnesium levels <2.0 mg/dL;
* Coexistent second malignancy or history of prior malignancy within previous 5 years (excluding basal or squamous cell carcinoma of the skin that has been treated curatively); or
* Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-05-07 (Actual); Primary Completion 2006-09-01 (Actual); Study Completion 2006-09-01 (Actual)

PRIMARY OUTCOMES:
Rate of objective disease control | Up to 6 months
  Rate of objective disease control was defined as the proportion of patients with confirmed CR, PR, or SD for at least 6 months, as determined by the Response Evaluation Criteria for Solid Tumors (RECIST).

REFERENCES:
- [Background] Molife LR, Attard G, Fong PC, Karavasilis V, Reid AH, Patterson S, Riggs CE Jr, Higano C, Stadler WM, McCulloch W, Dearnaley D, Parker C, de Bono JS. Phase II, two-stage, single-arm trial of the histone deacetylase inhibitor (HDACi) romidepsin in metastatic castration-resistant prostate cancer (CRPC). Ann Oncol. 2010 Jan;21(1):109-13. doi: 10.1093/annonc/mdp270. Epub 2009 Jul 16. PMID 19608618
- [Background] Rodon J, Perez-Fidalgo A, Krop IE, Burris H, Guerrero-Zotano A, Britten CD, Becerra C, Schellens J, Richards DA, Schuler M, Abu-Khalaf M, Johnson FM, Ranson M, Edenfield J, Silva AP, Hackl W, Quadt C, Demanse D, Duval V, Baselga J. Phase 1/1b dose escalation and expansion study of BEZ235, a dual PI3K/mTOR inhibitor, in patients with advanced solid tumors including patients with advanced breast cancer. Cancer Chemother Pharmacol. 2018 Aug;82(2):285-298. doi: 10.1007/s00280-018-3610-z. Epub 2018 Jun 7. PMID 29882016
- [Background] Barata PC, Cooney M, Mendiratta P, Tyler A, Dreicer R, Garcia JA. Ketoconazole plus Lenalidomide in patients with Castration-Resistant Prostate Cancer (CRPC): results of an open-label phase II study. Invest New Drugs. 2018 Dec;36(6):1085-1092. doi: 10.1007/s10637-018-0660-3. Epub 2018 Sep 6. PMID 30191523
- [Background] Komrokji RS, Al Ali NH, Padron E, Cogle C, Tinsley S, Sallman D, Lancet JE, Lis AF. Lenalidomide and Prednisone in Low and Intermediate-1 IPSS Risk, Non-Del(5q) Patients With Myelodysplastic Syndromes: Phase 2 Clinical Trial. Clin Lymphoma Myeloma Leuk. 2019 Apr;19(4):251-254. doi: 10.1016/j.clml.2018.12.014. Epub 2019 Jan 2. PMID 30852241
- [Background] Pal SK, Forero-Torres A, Thompson JA, Morris JC, Chhabra S, Hoimes CJ, Vogelzang NJ, Boyd T, Bergerot PG, Adashek JJ, Li H, Yu X, Gartner EM, Carret AS, Smith DC. A phase 1 trial of SGN-CD70A in patients with CD70-positive, metastatic renal cell carcinoma. Cancer. 2019 Apr 1;125(7):1124-1132. doi: 10.1002/cncr.31912. Epub 2019 Jan 9. PMID 30624766